## **RESEARCH CONSENT FORM**



## Improving medication adherence in kidney transplant patients; Can we help you to take your immunosuppressant medication?

| Na | ime of Principal Investigator: Dawn G | oodall | | |
|---|---|---|---|---|
| Th | is form documents your agreement to | o take part in this rese | | e initial box |
| 1. | I confirm that I have read and understand the participant information sheet dated 16 <sup>th</sup> January 2018 version 4 for the above study and have had the opportunity to ask questions which have been answered fully. | | | |
| 2. | I understand that my participation is voluntary and I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College Healthcare NHS Trust or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to access my records that are relevant to this research. | | | |
| 4. | I agree that all my study data, including identifiable data may be securely kept at Imperial College Healthcare NHS Trust for 5 years following completion of the study | | | |
| 5. | . I understand that once collected, my identifiable data and my contributions to the study will be retained and used in full, even if I become incapacitated. | | | |
| 6. | 6. I agree to my GP being informed of my participation in this study | | | |
| 7. | I agree to take part in the above study. | | | |
| If y | e you taking part in any other researd<br>your answer is yes, an assessment wi<br>appropriate to include you in this stu | ill be made by the res | search team in collaboration with you, whet | Yes / No<br>her it would |
| Na | me of participant | Signature | <br>Date | |
| Pa | rticipant's date of birth | | | |
| | ime of Person taking consent<br>different from Principal Investigator) | Signature | Date | |
| Pri | ncipal Investigator | Date | <br>Signature | |

V5.0 26/02/2018 IRAS Project ID 232623

1 copy for participant; 1 copy for Principal Investigator to scan into patient electronic record and then destroy.